CLINICAL TRIAL: NCT02168413
Title: Development of New Cortical Excitability Methodologies Using Robotised and Neuronavigated Transcranial Magnetic Stimulation.
Brief Title: Cortical Excitability Using Robotised and Neuronavigated Transcranial Magnetic Stimulation
Acronym: ROBEXCI
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A01734-41
Record Dates: First submitted 2014-05-23; First posted 2014-06-20 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2018-10

CONDITIONS: Cortical Excitability; Robotized TMS
Keywords: cortical excitability; robotized TMS; EEG; EMG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study has two main goals :

* to develop the cortcial excitbality (CE) measurement methodology using coupling between transcranial magnetic stimulation (TMS) and physiological recordings such as electroencephalography (EEG) and electromyography (EMG),
* to automatize these measurements using robotized TMS.

Assessing CE is a preliminary and crucial step in any TMS protocol, in either fundamental or clinical research. It is an important indicator which determine the stimulation power applied on the cortical target during the TMS experiment, or during the rTMS cure (patients). CE is in general measured on the motor cortex using EMG activity as the main indicator of the system's response, whatever the real cortical target is located. The present study thus propose to generalize this measurement on other cortical areas in link with the actual targets, and using other external recordings such as EEG. Moreover, as neuronavigation systems significantly improved TMS precision in the past years, CE measurements could significantly gain to become fully automatized using robotized TMS.

DETAILED DESCRIPTION:
Eligibility Criteria :

CRITERIA OF INCLUSION

* Major Topic (18 to 75)
* Signed informed consent,
* A medical examination must be done before participation in research,
* Membership or beneficiary of a social security scheme,

CRITERIA OF NON-INCLUSION

* Topic of under 18 and over 75 years.
* Against-indications (CI) to the practice of MRI pacemaker or implantable defibrillator or pacemaker neurosensory (risk of temporary or permanent damage to the device or heating metal parts). Cochlear implants (risk of demagnetization, electrode temperature rise and artifacts). Ocular or cerebral ferromagnetic foreign body close to the nerve structures (risk of displacement and complications such as eye or brain damage). Metal prostheses (possibility of significant artifacts according to their size and their ferromagnetic character, some neurosurgical clips or heart valves can cause problems and require an investigation into the exact model implanted). Topics claustrophobic. Pregnant woman. Neurosurgical ventriculoperitoneal bypass valves. Irremovable metal braces.
* CI practice of TMS: the history of epilepsy or seizures during hyperthermia during childhood are related ICs. Ferrométalliques body presence in the brain, cochlear implants, pacemakers, insulin pumps, during pregnancy, about jet lag or not having slept the night before the session of TMS.
* Existence of a severe condition in general terms: cardiac, respiratory, hematologic, renal, hepatic, cancerous,
* Regular Taking anxiolytics, sedatives, antidepressants, neuroleptics,
* Psychiatric disorder characterized,
* Alcohol ingestion before the examination,
* Persons referred to in Articles L1121-5 to L1121-8 CSP.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects (18 to 75 years old)
* consent form signed
* medical examination done prior to the experiment
* affiliated to the French social security

Exclusion Criteria:

* Exclusion criteria associated to MRI : pacemaker or neurosensory stimulator or implantable defibrillator. Cochlear implants. Ferromagnetic external bodies. Metal prosthesis. Claustrophobia. Pregnancy. Neurochirurgical bypass valves. Fixed metal dentures.
* Exclusion criteria associated to TMS : seizures antecedent. Pacemaker or neurosensory stimulator or implantable defibrillator. Cochlear implants. Ferromagnetic external bodies. Pregnancy. Insulin pump. Jet-lag or sleep deprivation. Severe medical affliction. Regular doses of anxiolytics, sedatives, antidepressant, neuroleptic. Psychiatric illness. Alcool ingestion prior to the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ealthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity (EMG) | One hour
  Participants' electromyographic activity will be recorded during an average of one hour.

SECONDARY OUTCOMES:
Electroencephalographic activity (EEG) | One hour
  Participants' electroencephalographic activity will be recorded during an average of one hour.

OTHER OUTCOMES:
Oculometry : saccadic eye movement | One hour
  Participants' saccadic eye movements will be recorded during an average of one hour.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry BOUGEROL, PUPH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- UMS CNRS 3552 IRMaGe, Grenoble, RA, France